CLINICAL TRIAL: NCT00708045
Title: A Multi-modality Imaging Assessment of Chemobrain
Acronym: Chemobrain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCI21946
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: [18F]fluoro-2-deoxy-D-glucose (FDG)

INTERVENTIONS:
Drug: [18F]fluoro-2-deoxy-D-glucose (FDG) — Brain scan with imaging tracer to assess brain tumor metabolism
  Other Names: FDG-PET; [18F]FDG; FDG-PET/CT

SUMMARY:
Patients must have had their breast cancer treated at the Huntsman Cancer Institute to be eligible for this trial.

OBJECTIVES:

To use quantitative FDG-positron emission tomography (PET), functional MRI (fMRI) and co-registered anatomic MRI imaging to better understand the cognitive disorder known as "chemobrain" which effects up to 16 -50% of individuals receiving long-term adjuvant chemotherapy [Tannock 2004, Matsuda 2005]. The study is exploratory to obtain proof of feasibility pilot data to support an eventual submission to the NIH.

Neuropsychological Testing A battery of testing will be used to assess the subjective complaints of cognitive impairment in the symptomatic patient cohort. Similarly the same battery of tests will be used to assure that the non-symptomatic patient control group and the age-matched normal controls do not exhibit any cognitive impairment. The following set of clinical tests will be performed to assess the degree of cognitive impairment in all subjects.

DETAILED DESCRIPTION:
In this study, 3 groups of 8 women each, between the ages of 18 and 65, will participate in this study. The "affected patient group" will be women with complaints of memory dysfunction who have received adjuvant chemotherapy (one or more anticancer drugs used in combination with surgery), for the treatment of breast cancer. These patients will be those that are being treated at Huntsman Cancer Institute/Hospital.

The second "patient control group" will be age-matched (same age) women with breast cancer who have undergone similar chemotherapy and have no complaints of memory problems.

The non-patient group will be age-matched (same age) women who have not undergone any type of chemotherapy. These individuals will be recruited from friends of female family members of the two breast cancer groups.

All individuals will be assessed for dementia (intellectual deterioration) and brain problems using the same kind of neuropsychological testing. All subjects will be age-matched as close as possible, to eliminate age related effects. Subjects will be right-handed, primarily-English speakers with normal hearing.

The purpose of this study is to use modern imaging techniques to better understand chemobrain. These imaging techniques include FDG-PET (FDG is the abbreviation for the radiopharmaceutical fluorodeoxyglucose and PET is Positron Emission Tomography) and functional MRI (fMRI)). They will be used to look at the metabolism (chemical activity) in specific areas of the brain and the entire brain overall. By using FDG-PET doctors will see how the brain activates. By using fMRI doctors will see how the brain works when you are challenged with certain mental tasks that make you concentrate and remember. FDG-PET and fMRI might provide important information on the brain that may be connected with chemotherapy.

This study will be an important first step to understand the problem of chemobrain. The imaging evaluations will make it possible to explore the changes in brain function that may be responsible for chemobrain and hopefully make it possible to predict which people may be affected by this problem.

Many people who undergo chemotherapy particularly adjuvant chemotherapy have complained about cognitive dysfunction for many years. This cognitive decline effects up to 16 -50% of individuals receiving long-term adjuvant chemotherapy [Tannock 2004, Matsuda 2005].Cancer survivors frequently refer to this cognitive dysfunction as "chemobrain" or "chemofog." The majority of individuals who are affected are woman who have undergone adjuvant chemotherapy for breast cancer. The table below is a summary of many of the studies that have been performed assessing cognition and chemobrain.

Women who experience chemobrain typically complain of inability to concentrate, memory dysfunction, word finding difficulties, difficulty with learning, slowed processing abilities, and often difficulty with writing and speaking. A particularly disturbing complaint for many individuals is the inability to multitask. Only recently, have researchers begun studying the impact of chemotherapy on cognitive functioning. This is a difficult area to study however. Part of the problem in assessing chemobrain using scientific principals is sorting out which problems are due to chemotherapy and which are due to having a serious illness like cancer that can result in physical debilitation, depression, sleep disruption, hormone shifts, and fatigue--all of which can affect cognitive functioning.

There are a number of theories at to why chemobrain may occur. One is that some types of chemotherapy can cross the blood/brain barrier and cause neurotoxicity. Another is that the cognitive problems are created by certain free radicals, the toxic elements that many types of chemotherapy produce [Joshi 2005]. Another theory is that some people have a genetic background that makes them more susceptible to the effects of chemotherapy. Most likely it is not just a single etiologic factor but a multifactorial process that combine to predispose certain individuals to develop chemobrain. Chemotherapy isn't the only cancer treatment that may cause cognitive disturbance and memory complaints. Other cancer treatments that have been implicated as causing complaints of cognitive dysfunction include hormone therapy, immunotherapy, and radiation therapy. Hormone therapy is common in woman being treated with conventional chemotherapy. It is not entirely clear if women undergoing hormone therapy which alters the amount of systemic estrogen experience memory problems. Some studies link memory to the amount of estrogen in the brain. Other studies haven't found this link.

ELIGIBILITY:
Inclusion criteria: Pre-screening will be conducted to ensure that all subjects are in good neurologic health with no history of seizures or other neurological disorders, and that they have no ferromagnetic implants or clips in their body. Subjects will be right-handed exclusive-English speakers with normal hearing.

Exclusion criteria: If a subject is found to have profound or severe depression after the Neuropsychological and Cognitive Testing session they may be excluded from the imaging portion of the study. This is justified as the imaging session would not be valid as the biologic correlates of depression rather than chemobrain would be imaged. Subjects found to have profound or severe depression will be notified and appropriate referral made to get them the necessary medical care to treat their depression.

Three cohorts of 8 women each under the age of 65 will be recruited for this exploratory pilot study. The "affected patient cohort" will be woman with complaints of cognitive or memory dysfunction who have received adjuvant chemotherapy for the treatment of breast cancer. These patients will be those being treated at Huntsman Cancer Hospital and be the patients of Dr Saundra Buys or Dr John Ward. The second "patient control cohort" will be age-matched woman with breast cancer who have undergone similar adjuvant chemotherapy for the same amount of time who have no complaints of memory dysfunction. Again these are primarily patients of Drs. Buys or Ward. The non-patient cohort will be age-matched woman who have not undergone any type of chemotherapy. These individuals will be recruited from friends of female family members of the two breast cancer cohorts. All individuals will be assessed for dementia and cognitive impairment using the same battery of dementia and cognitive/neuropsychological testing. All subjects will be age-matched as close as possible to eliminate age related cognitive effects. Subjects will be right-handed exclusive-English speakers with normal hearing. Pre-screening will be conducted to ensure that all subjects are in good neurologic health with no history of seizures or other neurological disorders, and that they have no ferromagnetic implants or clips in their body.

Up to 40 subjects may be enrolled to ensure 24 evaluable subjects.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-05-09 (Actual); Primary Completion 2015-02-05 (Actual); Study Completion 2015-02-05 (Actual)

PRIMARY OUTCOMES:
To use quantitative FDG-PET, functional MRI (fMRI) and co-registered anatomic MRI imaging to better understand the cognitive disorder known as "chemobrain" which effects up to 16 -50% of individuals receiving long-term adjuvant chemotherapy | December 2011
  To use quantitative FDG-PET, functional MRI (fMRI) and co-registered anatomic MRI imaging to better understand the cognitive disorder known as "chemobrain" which effects up to 16 -50% of individuals receiving long-term adjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yapp, PhD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States